CLINICAL TRIAL: NCT05991193
Title: A Non-interventional Study and Its Clinical Relevance With Central Nervous System Metastatic Epidermal Growth Factor Receptor Mutation Positive Non-small Cell Lung Cancer
Brief Title: A Study With Central Nervous System Metastatic EGFR Mutation Positive Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: FORCE RWS
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — needle biopsy for samples with DNA
Oversight: FDA-regulated Device: No

SUMMARY:
This is a descriptive observational study, in which data are collected in an epidemiological fashion and prospective. This study does not intend to intervene the current medical practice of the recruited patients.

DETAILED DESCRIPTION:
This is a descriptive observational study, in which data are collected in an EGFR mutant NSCLC. Our research plan aims to use multi-omics approaches to predict the likelihood of patients developing brain metastases, assess the prognosis of brain metastasis treatment, and identify potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years.
* Provision of fully informed consent prior to any study specific procedures.
* Patient with EGFR 19Del or L858R mutation diagnosed histologically or cytologically. The mutations above may exist alone or together.
* Patients must have untreated advanced Non-Small Cell Lung Cancer (NSCLC).
* According to the RECIST 1.1 standard, the patient must have at least one measurable lesion.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with EGFR 19Del or L858R mutation diagnosed histologically or cytologically.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression.

SECONDARY OUTCOMES:
Central nervous system (CNS) progression-free survival | 2 years
  CNS PFS is defined as the time from beginning of study treatment until the date of objective progression of central nervous system or death (by any cause in the absence of CNS progression), regardless of whether the patient withdraws from study treatment or receives another anti-cancer therapy prior to progression.
Objective Response Rate | 2 years
  Defined as the number (%) of patients with response of Complete Response or Partial Response

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China